CLINICAL TRIAL: NCT01705418
Title: Behavior Addictions Improvement in Parkinson Disease's Patients Treated by
Brief Title: Behavior Addictions Improvement in Parkinson Disease's Patients Treated by Subthalamic Stimulation : Long Term Follow-up
Acronym: PDdicted
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 12PHR02
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Deep brain stimulation; behavior and psychiatric symptoms improvement
MeSH Terms: conditions — Parkinson Disease; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Improvement of behavioral addictions in STN-DBS in PD: Long term follow-up

DETAILED DESCRIPTION:
Whereas subthalamic nucleus (STN) stimulation is considered an established treatment for motor symptoms in advanced Parkinson's disease (PD), its behavioral and psychiatric effects are strongly debated, with some studies showing a worsening or new onset of behavioral and psychiatric issues after STN stimulation and other showing an improvement. However, these data are based mainly on case reports and retrospective series.

Recently, the investigators group has conducted a prospective study assessing behavior and psychiatric symptoms in patients undergoing STN stimulation up to one year after surgery. After subthalamic stimulation non-motor fluctuations improved and pathologic hyperdopaminergic syndrome, i.e. behavioral addictions (including pathological gambling, hypersexuality, binge eating, compulsive shopping, …), compulsive use of dopaminergic treatment and dopaminergic dysregulation syndrome (defined as the association of one or more behavioral addictions to compulsive use of dopaminergic treatment), disappeared. These findings represent a milestone because, if confirmed, the indications of STN stimulation might be extended beyond motor complications. To date, there are several long-term studies on motor and cognitive effects of STN stimulation, whereas no long-term longitudinal data on neuropsychiatric effects do exist. Therefore, the investigators designed a long-term prospective study, assessing over 3-8 years behavioral and psychiatric effect in the same cohort of patients included in the one-year study. This study will allow to better evaluate the change in non-motor fluctuations and of behavioral issues in the long-term with a standard management.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the protocol 'Apathy'

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's desesase patients included in another protocol evaluating Apathy after deep brain stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbes M, Lhommee E, Thobois S, Klinger H, Schmitt E, Bichon A, Castrioto A, Xie J, Fraix V, Kistner A, Pelissier P, Seigneuret E, Chabardes S, Mertens P, Broussolle E, Moro E, Krack P. Subthalamic stimulation and neuropsychiatric symptoms in Parkinson's disease: results from a long-term follow-up cohort study. J Neurol Neurosurg Psychiatry. 2018 Aug;89(8):836-843. doi: 10.1136/jnnp-2017-316373. Epub 2018 Feb 7. PMID 29436490